CLINICAL TRIAL: NCT07233187
Title: The Effect of Continuous Wireless Fetal Monitoring During the Intrapartum Period on Labor Pain and Birth Experience: A Randomized Controlled Single-Blind Study
Brief Title: The Effect of Wireless Electronic Fetal Monitoring on Labor Pain and Birth Experiences
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Melek Şen Aytekin, Research Assistant Doctor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaU-EBE-MŞA-04
Record Dates: First submitted 2025-10-02; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Birth; Intrapartum
Keywords: Fetal Monitoring; intrapartum; pain; birth experience; Continuous Wireless Fetal Monitoring
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Wired EFM Group (No Intervention): In routine practice, fetal health assessments for pregnant women presenting for labor are conducted using a continuous wired EFM. Pregnant women in this group will not receive any interventions other than routine procedures. Because pregnant women are constantly connected to the EFM, the EFM will be removed and reconnected when necessary, such as when going to the toilet.
- Continuous Wireless EFM Group (Experimental): Pregnant women in this group will be continuously assessed with wireless EFM. Because it's a wireless application, pregnant women will have the freedom to move freely throughout labor. They will be able to perform their own activities, such as toileting, and other necessary activities. Pregnant women will not be subjected to any other procedures other than continuous wireless EFM.
  Interventions: Other: Continuous Wireless EFM Group

INTERVENTIONS:
Other: Continuous Wireless EFM Group — Pregnant women in this group will be continuously assessed with wireless EFM. Because it's a wireless application, pregnant women will have the freedom to move freely throughout labor. They will be able to perform their own activities, such as toileting, and other necessary activities. Pregnant women will not be subjected to any other procedures other than continuous wireless EFM.
  Arms: Continuous Wireless EFM Group

SUMMARY:
This study is using Electronic Fetal Monitoring (EFM) to assess fetal health in pregnant women in labor. This will be compared with continuous wired EFM and continuous wireless EFM. The effects of wireless and continuous wireless EFM on labor pain levels and labor experiences will be measured.

DETAILED DESCRIPTION:
In this study, Electronic Fetal Monitoring (EFM) is being applied to pregnant women in labor to assess fetal health. This procedure is typically performed in hospitals using a continuous wired EFM. During this period, women are forced to lie down constantly and cannot use active methods to cope with pain. Therefore, using a wireless EFM may be an approach that allows for continuous assessment while also supporting women's activity. Therefore, a comparison will be made between continuous wired EFM and continuous wireless EFM. During labor, pain levels will be assessed using the Visual Analog Scale when cervical dilation is between 8 and 10 cm. After the first hour postpartum, the labor experience of the postpartum woman will be collected using the Birth Experiences Scale.

ELIGIBILITY:
Inclusion Criteria:

* The study included healthy primiparous or multiparous pregnant women who agreed to participate in the study, were between the ages of 18 and 35, had a gestational age greater than 37+0, had cervical dilation greater than 4 cm, had a single, live fetus, were not using uterotonic agents, spoke Turkish, had no comprehension, perception, or communication problems, and were healthy.

Exclusion Criteria:

* Pregnant women who were diagnosed with a risky pregnancy, who were illiterate, who had a contagious disease, or who had a risky disease were not included in the study.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since the study will be conducted with pregnant women in the intrapartum period, only women will be biologically eligible to be included in the study.
Enrollment: 112 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Birth Experience Questionnaire | 1 hour after the end of labor
  The Birth Experience Questionnaire (CEQ), developed by Dencker and colleagues in 2010, was adapted into Turkish by Mamuk and colleagues in 2019. Developed to measure women's birth experiences across various dimensions, the scale has four subscales and 22 items. It consists of the following subscales: Birth Process (8 items), Professional Assistance/Support (5 items), Perceived Safety/Memories (6 items), and Participation in Decisions (3 items).
The Visual Acuity Scale | Determining the pain level of pregnant women will be completed within 5 minutes when cervical dilation is 8-10 cm.
  This is a horizontal or vertical line, usually 10 cm long, used to assess pain intensity. It begins with "No Pain" and ends with "Unbearable Pain." The patient marks the appropriate location on this line based on the pain they experience. The VAS is used to convert some values that cannot be measured numerically into numerical values. The two extremes of the parameter to be evaluated are written at either end of a 100 mm line, and the patient is asked to indicate where their own condition aligns with this line by drawing a line, placing a dot, or pointing. For example, for pain, "No pain at all" is written at one end, and "Extreme pain at the other end," and the patient marks their current condition on this line. According to this scale, the patient is asked to rate whether they have pain or not, and if so, to rate it on a scale of 0-10. According to this score, pain intensity is considered mild pain at <3, moderate pain at 3-6, and severe pain at >6. The distance from the point of

SECONDARY OUTCOMES:
Personal Information Form | The data will be collected 5 minutes after the pregnant woman is included in the study.
  This form, which questions the introductory characteristics of pregnant women, consists of a total of 23 questions, 6 of which are to determine the socio-demographic and obstetric characteristics of pregnant women, 8 questions to learn their obstetric information and 9 questions about birth experience.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Şen Aytekin, Research Assistant, Principal Investigator — Tokat Gaziosmanpasa University; Demet Çakır, Assistant Professor, Study Chair — Tokat Gaziosmanpasa University; Ayşenur Kahraman, Research Assistant, Study Chair — Tokat Gaziosmanpasa University; Emine Aksüt Akçay, Study Chair — Kahramanmaras Sütcü İmam Unıversity
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No